CLINICAL TRIAL: NCT03018860
Title: Alternative to Intensive Management of the Active Phase of the Second Stage of Labor : a Multicenter Randomized Controlled Trial
Brief Title: Alternative to Intensive Management of the Active Phase of the Second Stage of Labor
Acronym: PASST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P150937
Record Dates: First submitted 2017-01-03; First posted 2017-01-12 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Active Second Stage
Keywords: Active second stage; Neonatal morbidity; Operative delivery; Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Moderate" management (Experimental): Women are encouraged by physicians to push only 2 times per contractions, to respect contractions without pushing and there is no limit of pushing duration.
  Interventions: Procedure: "Moderate" management
- "Intensive" management (Active Comparator): Usual obstetrical care in France
  Interventions: Procedure: "Intensive" management

INTERVENTIONS:
Procedure: "Moderate" management — After randomization, women allocated to the intervention group, i.e. "moderate" pushing, are encouraged to push only 2 times per contractions, to respect contractions without pushing and there is no limit of pushing duration.
  Arms: "Moderate" management
Procedure: "Intensive" management — This group corresponds to usual obstetrical management of active second stage in France. In France, national guidelines recommend to limit maternal expulsive efforts to 30 minutes (grade C). Thus, physicians (midwives and obstetricians) encourage usually women to push 3 times per contractions and to push on every contraction in order to deliver into a 30 minutes timing.
  Arms: "Intensive" management

SUMMARY:
Active phase of the second stage of labor corresponds to period of maternal expulsive efforts (i.e. pushing). An intensive management of this phase is usual in France. This study aims to evaluate the impact of an alternative "moderate" management during this pushing phase on neonatal and maternal issues and mode of delivery.

DETAILED DESCRIPTION:
Management of the active phase of the second stage of labor is not an evidence-based practice. Management of this phase differs between countries. In France, national guidelines recommend to limit maternal expulsive efforts to 30 minutes (grade C). Thus, physicians (midwives and obstetricians) encourage usually women to push 3 times per contractions and to push on every contraction in order to deliver into a 30 minutes timing.

This study aims to evaluate the impact of an alternative "moderate" management during this pushing phase on neonatal and maternal issues and mode of delivery. In the intervention group, i.e. "moderate" pushing, women are encouraged to push only 2 times per contractions, to respect contractions without pushing and there is no limit of pushing duration.

The hypothesis is that "moderate" management of the active phase of the second stage allows decreasing frequency of neonatal morbidity at birth, decreasing frequency of operative delivery and increasing maternal satisfaction.

ELIGIBILITY:
Inclusion Criteria :

* primiparous women
* singleton fetus
* fetal cephalic presentation
* ≥37 gestational weeks
* living fetus
* Patient with epidural analgesia
* Major Female
* Women understand French

Exclusion Criteria :

* Abnormal fetal heart rate requiring hastening childbirth
* cervical dilatation < 8 cm
* intrauterine fetal growth restriction <5e percentile,
* Fetal malformation,
* history of gynecological surgery with uterine scar
* Women do not understand French,
* women with psychiatric condition
* contraindication to intensive management of active second stage (severe myopia, respiratory or cardiac failure)
* no affiliation to a social security scheme (beneficiary or assignee)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1701 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Neonatal morbidity composite measure | at childbirth
  number of participant with acidosis arterial cord pH <7.15 and / or excess base> 10 mmol / L and / or lactate> 6 mmol / L and or an Apgar score at 5 minutes <7 and or severe neonatal trauma defined by fractures, brachial plexus, facial paralysis, cephalohematoma, intracerebral hematoma other (neonatal morbidity composite measure) and or an Apgar score at 5 minutes <7 and or severe neonatal trauma: fractures, brachial plexus, facial paralysis, cephalohematoma, intracerebral hematoma other (neonatal morbidity composite measure)

SECONDARY OUTCOMES:
Mode of delivery | at childbirth
  spontaneous vaginal, instrumental vaginal delivery or cesarean section
Immediate postpartum complications | 2 hours after delivery
  Perineal lesions with involvement of the anal sphincter (3rd and 4th degree)
Immediate postpartum complications | 2 hours after delivery
  Episiotomy
Immediate postpartum complications | 2 hours after delivery
  Cervical and vaginal lesion
Immediate postpartum complications | 2 hours after delivery
  Severe postpartum hemorrhage (blood loss estimated> 1000 mL, using sulprostone, intrauterine bloating, transfusion, uterine artery embolization, vessel ligation, uterine upholstery, of hysterectomy)
Immediate postpartum complications | 2 hours after delivery
  Postpartum Hemorrhage (blood loss estimated> 500mLand < 1000mL)
Women satisfaction assessed with the Labour Agentry scale | 2 hours after delivery
Women satisfaction assessed with the ICIQ-UI Short Form | 6 months post partum
Urinary and anal incontinence assessed with the Wexner Score | 6 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves ANCEL, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Ray C, Rozenberg P, Kayem G, Harvey T, Sibiude J, Doret M, Parant O, Fuchs F, Vardon D, Azria E, Senat MV, Ceccaldi PF, Seco A, Garabedian C, Chantry AA; Groupe de Recherche en Obstetrique et Gynecologie. Alternative to intensive management of the active phase of the second stage of labor: a multicenter randomized trial (Phase Active du Second STade trial) among nulliparous women with an epidural. Am J Obstet Gynecol. 2022 Oct;227(4):639.e1-639.e15. doi: 10.1016/j.ajog.2022.07.025. Epub 2022 Jul 19. PMID 35868416
- [Background] Le Ray C, Audibert F. [Duration of pushing in labor: literature review]. J Gynecol Obstet Biol Reprod (Paris). 2008 Jun;37(4):325-8. doi: 10.1016/j.jgyn.2008.02.009. Epub 2008 Apr 10. French. PMID 18406074
- [Background] Nordstrom L, Achanna S, Naka K, Arulkumaran S. Fetal and maternal lactate increase during active second stage of labour. BJOG. 2001 Mar;108(3):263-8. doi: 10.1111/j.1471-0528.2001.00034.x. PMID 11281466
- [Background] Le Ray C, Audibert F, Goffinet F, Fraser W. When to stop pushing: effects of duration of second-stage expulsion efforts on maternal and neonatal outcomes in nulliparous women with epidural analgesia. Am J Obstet Gynecol. 2009 Oct;201(4):361.e1-7. doi: 10.1016/j.ajog.2009.08.002. PMID 19788968
- [Background] Cheng YW, Hopkins LM, Caughey AB. How long is too long: Does a prolonged second stage of labor in nulliparous women affect maternal and neonatal outcomes? Am J Obstet Gynecol. 2004 Sep;191(3):933-8. doi: 10.1016/j.ajog.2004.05.044. PMID 15467567
- [Background] Dionne MD, Deneux-Tharaux C, Dupont C, Basso O, Rudigoz RC, Bouvier-Colle MH, Le Ray C. Duration of Expulsive Efforts and Risk of Postpartum Hemorrhage in Nulliparous Women: A Population-Based Study. PLoS One. 2015 Nov 10;10(11):e0142171. doi: 10.1371/journal.pone.0142171. eCollection 2015. PMID 26555447
- [Derived] Dupuis N, Pizzoferrato AC, Garabedian C, Rozenberg P, Kayem G, Harvey T, Mandelbrot L, Doret M, Fuchs F, Azria E, Senat MV, Ceccaldi PF, Seco A, Chantry A, Le Ray C; GROG (Groupe de Recherche en Obstetrique et Gynecologie). Moderate or intensive management of the active phase of second-stage labor and risk of urinary and anal incontinence: results of the PASST randomized controlled trial. Am J Obstet Gynecol. 2023 Nov;229(5):528.e1-528.e17. doi: 10.1016/j.ajog.2023.07.034. Epub 2023 Jul 26. PMID 37499991